CLINICAL TRIAL: NCT07268079
Title: Validation Study of VIRADIA: A Virtual Reality Diagnostic Platform for the Assessment of Neurological and Cognitive Functions
Brief Title: Validation of the VIRADIA App for Neurological and Cognitive Diagnostics in Virtual Reality
Acronym: VIRADIA
Status: Recruiting | Type: Observational
Sponsor: Gametherapy (Other)
Responsible Party: Sponsor
Other Study IDs: 09I05-03-V04; 09I05-03-V04 (Other: Local Ethics Committee NSK Slovakia)
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Neurological Disorders; Cognitive Impairment; Motor Impairment; Neurodegenerative Diseases
Keywords: Virtual Reality; Neurological Diagnostics; Cognitive Assessment; Motor Function; Neuropsychology; Validity; Digital Health
MeSH Terms: conditions — Nervous System Diseases; Cognitive Dysfunction; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: Healthy adult volunteers without known neurological or psychiatric conditions. Participants complete both the standard (paper-based or face-to-face) and Virtual Reality (VR) versions of all diagnostic tests.
  Interventions: Diagnostic Test: VIRADIA - Virtual Reality Diagnostic Platform
- Neurological Patients: Adults with a confirmed neurological diagnosis (e.g., Parkinson's disease or related motor/cognitive disorder). Participants complete both the standard and Virtual Reality versions of the diagnostic tests.
  Interventions: Diagnostic Test: VIRADIA - Virtual Reality Diagnostic Platform

INTERVENTIONS:
Diagnostic Test: VIRADIA - Virtual Reality Diagnostic Platform — Participants complete a series of diagnostic tests in the VIRADIA virtual reality environment.

SUMMARY:
The VIRADIA study aims to validate and assess the reliability of a newly developed Virtual Reality (VR) diagnostic platform designed for neurological and cognitive testing. The goal is to determine whether the VR versions of nine commonly used clinical tests measure the same constructs and provide comparable results to their traditional face-to-face or paper-based forms.

The study includes two groups of participants: (1) healthy volunteers and (2) patients with neurological diagnoses. Each participant will complete both the standard and the VR versions of the tests, with the order of administration randomly assigned. The tested functions cover fine motor skills, gait and balance, attention, executive function, processing speed, and visuospatial abilities.

The following tests are included in the VR platform: 9-Hole Peg Test (9HPT), 6 Meter Walk Test, Timed Up and Go - Manual (TUG-M), Functional Reach Test (FRT), Symbol Digit Modalities Test (SDMT), Clock Drawing Test (CDT), Trail Making Test (TMT A/B), Stroop Test, and SATURN Test.

Participants will first provide informed consent and basic demographic information. They will then complete all tests in both modalities (standard and VR), with appropriate breaks between tasks.

The study is observational, within-subjects, and paired in design. Primary outcomes include correlation and agreement between VR and standard test scores (validity). Data will be analyzed using paired statistical methods, including Pearson/Spearman correlations, Bland-Altman analysis, and Intraclass Correlation Coefficients (ICC).

No medication or invasive intervention is used in this study. The VR testing is non-invasive and carries minimal risk. The study has been approved by the Ethics Committee of the Nitra Self-Governing Region (Approval No. 09I05-03-804).

The results will provide evidence for the validity and reliability of VR-based diagnostics and support the use of the VIRADIA platform as a safe, standardized tool for neurological and cognitive assessment.

DETAILED DESCRIPTION:
The VIRADIA validation study investigates the psychometric properties-validity and reliability-of a Virtual Reality (VR) diagnostic platform designed for neurological and cognitive assessment. The platform includes VR adaptations of nine established clinical tests commonly used in neurology and neuropsychology. These tests evaluate fine motor coordination, gait and balance, processing speed, attention, and executive functioning.

The study follows an observational, within-subjects, paired design. Each participant completes both the standard (paper-based or face-to-face) version and the corresponding VR version of all tests. The order of modalities is counterbalanced across participants to control for order effects. Two groups are enrolled:

1. Healthy adults (control group)
2. Patients with neurological conditions (clinical group; one priority diagnosis in the first phase)

Objectives

1. To evaluate the convergent validity of VR-based test scores compared to standard clinical versions.
2. To analyze discriminative validity, i.e., whether VR test results can differentiate between healthy individuals and neurological patients comparably to standard methods.

Procedures

After informed consent, demographic and clinical data (age, gender, education, diagnosis, medication) are recorded. Participants complete all tests under both conditions (standard and VR). After testing, participants fill out a short questionnaire on VR tolerability and subjective experience.

Data Collection and Sample Size

The study aims to include 200 participants (100 healthy, 100 patients). The target sample size was determined using a priori power analysis for paired ROC/AUC comparisons (AUC ≥ 0.75, ΔAUC ≤ 0.05, α = 0.05, power = 0.90), with an additional 15% margin for attrition.

Statistical Analyses

1. Convergent validity: Pearson/Spearman correlations (95% CI) between VR and standard scores.
2. Agreement: Paired t-tests/Wilcoxon tests and Bland-Altman plots (bias, 95% limits of agreement).
3. Discriminative validity: ROC/AUC analysis comparing patients and healthy participants.
4. Reliability: Intraclass Correlation Coefficient (ICC[2,1]) for the test-retest subsample.

Ethical Considerations

The study is non-invasive and presents minimal risk. No experimental drug, device, or biological material is used. All participants provide informed consent prior to participation. The study has been approved by the Ethics Committee of the Nitra Self-Governing Region (Approval No. 09I05-03-804).

Expected Outcomes

The study will produce empirical evidence supporting the validity, reliability, and clinical utility of the VIRADIA platform. This validation will enable the integration of standardized VR-based diagnostics into neurological practice and contribute to early detection of neurodegenerative disorders in both clinical and home settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Ability to provide informed consent.
* Adequate vision and hearing to complete testing.
* For the neurological group: confirmed diagnosis of a neurological disorder (e.g., Parkinson's disease, multiple sclerosis, or similar).
* For the control group: no history of neurological or psychiatric disease.

Exclusion Criteria:

* Severe cognitive impairment (MMSE < 24 or equivalent clinical judgment).
* Acute neurological or psychiatric condition interfering with testing.
* Severe motor disability preventing task performance (e.g., inability to use VR controller).
* Current substance abuse.
* Uncorrected visual impairment or vestibular disorder leading to intolerance of VR.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-80 years, including healthy volunteers and patients with neurological diagnoses recruited from outpatient neurology clinics and community sources in Nitra, Slovakia. Participants are screened for eligibility, provide informed consent, and complete both standard and Virtual Reality versions of diagnostic tests.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Virtual Reality (VR) and Standard Test Scores | Single assessment on Day 1 (one testing session)
  Convergent validity will be assessed by correlating participants' performance on the VR versions of nine diagnostic tests (9HPT, 25FWT, TUG-M, FRT, SDMT, CDT, TMT-A/B, Stroop, and SATURN) with their corresponding standard (paper or face-to-face) versions.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Menkyova, MD, PhD., Principal Investigator; Martin Polak, Dr., Principal Investigator — Gametherapy
Locations (1):
- INNER s.r.o., Fatranská 873/12, 94901 Nitra, Nitra, Nitra Region, Slovakia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive clinical and neurological information collected under local ethics approval for internal validation purposes only. Aggregate data and statistical results will be published in peer-reviewed journals.

REFERENCES:
- See also: Related Info — https://gametherapy.eu/viradia-diagnostic-platform

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT07268079/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT07268079/ICF_001.pdf